CLINICAL TRIAL: NCT02169622
Title: A Prospective Look at Incidence of Atrial Fibrillation After Coronary Artery Bypass Graft and Related Morbidity/Mortality Utilizing the Reveal XT
Brief Title: CABG REVEAL: Atrial Fibrillation After Coronary Artery Bypass Graft
Status: Completed | Type: Observational
Sponsor: Saint Thomas Health (Other)
Responsible Party: Sponsor
Other Study IDs: STH12-009; STH12-009 (Other: Saint Thomas Health)
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial Fibrillation is an abnormal heart rhythm that can occur after coronary heart bypass graft operations. How often this happens and what other problems occur for a person after these operations needs to be better understood. This study uses a device called the Reveal XT, a small device that records heart rhythms to track a patient's heart rhythms after the bypass surgery. The device is implanted at the time the bypass graft is made. The information that is gathered for this study will help physicians to provide better treatment and follow-up of the patients under their care.

DETAILED DESCRIPTION:
We will utilize the Reveal XT implantable loop recorder (ILR) in order to monitor the incidence of AF in our post-CABG patients. The Reveal XT has been shown to be superior in comparison to the more commonly used sporadic ECGs.6 Unfortunately, the occurrences of arrhythmias tend to be "unpredictable" and often paroxysmal. Observers are unlikely to have the opportunity to record ECGs at the time of event until it is too late. The ability of the Reveal XT to continuously record ECGs over long periods of time has made it a superior and powerful diagnostic tool in patients with arrhythmias and arrhythmia related complications.

This was evident in the large multicenter PICTURE study whereby a large number of diagnostic tests were undertaken in patients with unexplained syncope without providing conclusive data, but in the same study with the Reveal ILR, the mechanism of syncope in the vast majority of these patients were established often at first onset of an arrhythmia.7

"The equivalent efficacy", if not superiority, of Reveal ILRs above conventional ECGs and Holter-monitors in detecting AF was established in the "XPECT" trial.8 Its sensitivity in detecting events not seen with ECGs and Holter monitoring post COX MAZE procedure (surgical procedure for AF) and post ablations for paroxysmal AF and persistent AF is well established.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Presenting for elective Coronary Artery Bypass Graft at Saint Thomas West Hospital

Exclusion Criteria:

* Patients <60 years of age
* Prior cardiac surgery
* Emergent surgery
* Need for concomitant cardiac surgery other than PFO closure
* Prior history of AF or Atrial flutter
* Prior atrial ablation
* Prior cardioversion
* Patients with prior permanent pacemaker
* Ejection fraction <35%
* Prior history of thyroid disease
* Prior history of a cardiomyopathy
* Patients without telephonic access

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 60 years of age or older undergoing coronary artery bypass grafting (CABG).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Number and cost of atrial fibrillation after coronary artery bypass grafting (CABG) per patient | Three year follow-up
  Patient follow up
Number of complication s related to atrial fibrillation in patients after CABG | 3 year follow up
  Patient follow up
Number of therapeutic/intervention changes for participants post CABG resulting from use | 3 year follow up
  Patient follow up

CONTACTS AND LOCATIONS:
Overall Officials: Evelio Rodriquez, MD, Principal Investigator — Saint Thomas Heart at Saint Thomas
Locations (1):
- Saint Thomas West Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No